CLINICAL TRIAL: NCT00373425
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Single-agent Tarceva® (Erlotinib) Following Complete Tumor Resection With or Without Adjuvant Chemotherapy in Patients With Stage IB-IIIA Non-small Cell Lung Carcinoma Who Have EGFR-positive Tumors
Brief Title: A Study of Erlotinib (Tarceva) After Surgery With or Without Adjuvant Chemotherapy in Non-Small Cell Lung Carcinoma (NSCLC) Patients Who Have Epidermal Growth Factor Receptor (EGFR) Positive Tumors
Acronym: RADIANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSI-774-302; 2005-001747-29 (EudraCT Number)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Adjuvant Non-small Cell Lung Cancer; Tarceva; Early-stage Lung Cancer; Adjuvant; RADIANT; NSCLC; EGFR-positive tumor; Stage IB Non-small Cell Lung Cancer; Stage II Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib (Experimental): Participants received 150 mg/day erlotinib orally for 2 years or until relapse, death, participant request or investigator decision to discontinue study drug, or intolerable toxicity.
  Interventions: Drug: Erlotinib
- Placebo (Placebo Comparator): Participants received matching placebo tablets orally for 2 years or until relapse, death, participant request or investigator decision to discontinue study drug, or intolerable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — 150 mg tablet
  Other Names: OSI-774; Tarceva
  Arms: Erlotinib
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
This is a study to evaluate the effectiveness of erlotinib compared with a placebo sugar pill following complete surgical removal of the tumor with or without chemotherapy after surgery in Stage IB-IIIA NSCLC patients.

DETAILED DESCRIPTION:
After the initiation of the study, the sponsor became aware of an error in the drug dispensing module of the interactive voice response such that most patients who were randomized prior to 07 November 2007 were dispensed the incorrect study drug at least once. Since the integrity of the data from these patients was seriously compromised, these patients were considered unevaluable for the protocol-specified analyses. These participants are referred to as the breached protocol cohort (BPC) and those still on study treatment at the time of the breach were offered the option of receiving open-label erlotinib for up to 2 years (including posttreatment and long-term follow-up assessments), not receiving open-label erlotinib but remaining in the study for posttreatment and long-term follow-up assessment, or withdrawing consent from treatment and further assessments. Participants who had discontinued study treatment prior to the breach were not offered open-label erlotinib and remained in long-term follow-up. Data from the BPC participants were analyzed separately and were not included in the assessments of primary or secondary endpoints in the randomized cohort and were not considered part of the primary analyses.The sample size for the randomized cohort was not changed due to the BPC and the data from RC and BPC were analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Primary tissue from patient's surgery must be epidermal growth factor receptor (EGFR)-positive by certain tests
* Patients may have up to 4 cycles of chemotherapy after surgery
* Complete removal of the tumor by surgery
* Able to start drug under the following timelines:

  * 6 months from the day of surgery for patients who get chemotherapy
  * 3 months from the day of surgery for those who do not get chemotherapy
* Confirmed diagnosis of Stage IB-IIIA NSCLC
* Patients must be accessible for follow-up visits

Exclusion Criteria:

* History of prior radiotherapy for NSCLC either before or after surgery
* History of heart disease or uncontrolled heart arrhythmias within the previous year
* History of poorly controlled gastrointestinal (GI) disorders that could affect the absorption of study drug
* History of other cancer except certain skin or cervical cancers, patients who have had other cancer are eligible if they have remained disease free for at least 5 years
* Patients who have received chemotherapy for NSCLC before surgery
* Tumors with mixed histology of NSCLC and Small Cell Lung Cancer (SCLC). Patients with carcinoid tumors are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2006-09; Primary Completion 2013-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (285):
- United States (139):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Nat'l Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - USC/ Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - University of California, San Francisco Comprehensive Cancer Center, San Francisco, California
  - City of Hope Medical Group (COHMG), South Pasadena, California
  - Rocky Mountain Cancer Center- Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose St. Francis Health Services, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers- Rose, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Center-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Center-Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center, Sharon, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Smilow Cancer Hospital Care Center, Torrington, Connecticut
  - Florida Cancer Institute-New Hope, Hudson, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Watson Clinic LLP, Lakeland, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Institute- New Hope, New Port Richey, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Peachtree Hematology-Oncology Consultants, P.C., Atlanta, Georgia
  - Central Georgia Cancer Care, PC, Macon, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Mountain States Tumor Institute, Boise, Idaho
  - Mountain States Tumor Institute, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Mountain States Tumor Institute, Twin Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Section of Hematology/Oncology, Chicago, Illinois
  - Joliet Oncology Hematology Assoc., LTD, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health, Carmel, Indiana
  - Indiana University Health, Fishers, Indiana
  - Indiana University Health, Greenfield, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Cancer Care of Maine, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - St. Joseph Medical Center's Cancer Institute, Towson, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A., Burnsville, Minnesota
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Oncology Hematology, Saint Paul, Minnesota
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Heartland Regional Medical Center d/b/a Heartland Clinic, Saint Joseph, Missouri
  - St. Francis Cancer Treatment Center, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NH Oncology-Hematology PA (Co), Concord, New Hampshire
  - NH Oncology-Hematology PA, Hooksett, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Interlakes Oncology Hematology, PC, Brockport, New York
  - Interlakes Oncology Hematology, PC, Canadaigua, New York
  - Interlakes Oncology Hematology, PC, Geneva, New York
  - Advanced Oncology Associates, New Rochelle, New York
  - The New York Presbyterian-Weill Medical College of Cornell University, New York, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Raleigh Hematology Oncology Associates d/b/a Cancer Center of North Carolina, Cary, North Carolina
  - Carolina Oncology Specialists PA, Hickory, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Aultman Hospital/ North Canton Medical Foundation, Canton, Ohio
  - University Hopsitals of Cleveland, Cleveland, Ohio
  - Hematology Oncology Consultants Inc., Columbus, Ohio
  - Earle A Chiles Research Institute, Portland, Oregon
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Cancer Care Associates - Medical Oncology, Bethlehem, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - South Carolina Oncology Assoc., PA, Columbia, South Carolina
  - Cancer Centers of the Carolinas, Easley, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas, Spartanburg, South Carolina
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Bostin Baskin Cancer Foundation, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Bostin Baskin Cancer Foundation, Memphis, Tennessee
  - Family Cancer Center Foundation, Inc., Memphis, Tennessee
  - West Clinic, Memphis, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, P.A. - Amarillo, Amarillo, Texas
  - Texas Oncology Beaumont, Beaumont, Texas
  - Texas Oncology Texas Cancer Center at Medical City, Dallas, Texas
  - Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Flower Mound, Flower Mound, Texas
  - Texas Oncology, Fort Worth, Fort Worth, Texas
  - Texas Oncology Southwest Forth Worth, Fort Worth, Texas
  - Texas Oncology, Garland, Garland, Texas
  - Cancer Care Centers of South Texas - HOAST, New Braunfels, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Cancer Care Centers of South Texas-HOAST, San Antonio, Texas
  - Texas Oncology -Tyler, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Onc and Hem Associates of SW VA, Inc. d/b/a Blue Ridge Cancer Care, Christiansburg, Virginia
  - Onc and Hem Associates of SW VA, Inc., Christiansburg, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc. d/b/a Blue Ridge Cancer Care, Roanoke, Virginia
  - Onc and Hem Assoc of SW VA, Inc d/b/a Blue Ridge Cancer Care, Salem, Virginia
  - Onc and Hem Associates of SW VA, Inc. d/b/a Blue Ridge Cancer Care, Wytheville, Virginia
  - Univ. of Washington/ Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Cancer Care Northwest-North, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane Valley, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Northwest Cancer Specialist, P.C., Vancouver, Washington
- Argentina (5):
  - COIR, Mendoza, Mendoza Province
  - ISIS Centro Especializado De Luce S.A., Santa Fé, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Rehabilitación Respiratoria María Ferrer, Buenos Aires
  - Hospital Espanol de Rosario, Rosario, Santa Fe
- Australia (8):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Monash Medical Centre, East Bentleigh, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Respiratory Clinical Trials Pty., Ltd, Adelaide
  - Ashford Cancer Centre, Ashford
- Austria (7):
  - Universitaetsklinikum Innsbruck, Innsbruck
  - Allgemeines Krankenhaus der Stadt Linz, Linz
  - Landeskrankenhaus SalzburgUniversitaetsklinikum der PMUUniversitaetsklinik für Pneumologie, Salzburg
  - AKH Wien, Vienna
  - Krankenhaus Hietzing, Vienna
  - SMZ Baumgartner Hoehe - Otto Wagner Spital, Vienna
  - SMZ Baumgartner Höhe - Otto- Wagner-Spital, Vienna
- Belgium (4):
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Le Grand Hôpital de Charleroi, Charleroi
  - Centre Hospitalier Jolimont-Lobbes, La Louvière
- Canada (12):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Center of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional cancer Centre at Southlake, Newmarket, Ontario
  - RS MacLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill Dept. of Oncology, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - St. Joseph's Health Centre, Toronto
- Czechia (3):
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Fakultni nemocnice OstravaKlinika tuberkulozy a respiracnich nemoci, Ostrava-Poruba
  - FN Bulovka Klinika plincni a hrrudni chirurgie, Prague
- France (13):
  - CHU Larrey Service de Pneumologie, Clinique des voies respiratoires, Toulouse, Cedex 9
  - Centre d'Oncologie et de Radiothérapie du Pays Basque, Bayonne
  - C.H.U. Morvan, Institut de Cancerologie et d'Hématologie, Brest
  - CHU de Caen - Service de pneumologie, Caen
  - CHU Clermont Ferrand - Hôpital Gabriel Montpied - Service de pneumologie, Clermont-Ferrand
  - Hopital De La Croix-Rousse Service de Pneumologie, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital de Tenon, Paris
  - Fondation Hôpital Saint Joseph, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - CHU - Hopital Pontchaillou - Service de pneumologie, Rennes
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (19):
  - Zentralklinik Bad Berka, Bad Berka
  - HELIOS Klinikum Emil von Behring GmbH, Berlin
  - Augusta-Krankenanstalt Bochum, Bochum
  - Fachkrankenhaus Coswig, Coswig
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Göttingen, Göttingen
  - Lungenclinic Großhansdorf, Großhansdorf
  - Städtisches Krankenhaus Martha-Maria, Halle-Dölau, Halle
  - Asklepios Klinik Harburg, Hamburg
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklink Hemer des Deutschen Gemeinschafts-Diakonieverbandes GmbH, Hemer
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Mainz, Mainz
  - Asklepios Klinikum Gauting, Muenchen-Gauting
  - Pius Hospital Oldenburg, Oldenburg
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
- Greece (3):
  - IASO GENERAL Hospital of Athens, Athens
  - "Papageorgiou" General Hospital of Thessaloniki, Thessaloniki
  - "G. Papanikolaou" General Hospital of Thessaloniki, Thessaloniki
- Hungary (6):
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar Pulmonologiai Klinika, Budapest
  - Csongrad Megyei Onkormanyzat, Mellkasi Betegsegek Szakkorhaza, Deszk
  - Pecsi Tudomany Egyete m Klinikai Kozpont, I.sz Belgyogyaszati Klinika Pulmonologiai Munkacsoport, Pécs
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Vas Megyei Markusovszky Lajos Altalanos Rehabilitacios es Gyogyfurdo Korhaz, Egyetemi Oktatoko Zarkoruen Mukodo Nonprofit Reszveny Tarsasag, Szombathely
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I, Ancona
  - Ospedale Bellaria, Bologna
  - Ospedale Garibaldi Nesima, Catania
  - Istituto Nazionale per la Ricerca e la Cura del Cancro, Genova
  - Azienda Ospedaliero- Universitaria di Parma, Parma
  - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
- Poland (6):
  - Samodzielny Publiczny Szpital Kliniczny Nr 4, Lublin
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkoposkie Centrum Pulmonologii i Torakochirurgii, Oddzial Onkologii Klinicznej z Pododdzialem Dziennej Chemioterapii, Poznan
  - Specjalistyczny Szpital im. prof.Alfreda Sokolowskiego, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skllodowskiej - Curie, Warsaw
  - Dolnoslaskie Centrum Chorob Pluc we Wroclawiu, Katedra i Klinika Pulmonologii i Nowotworow Pluc Akademii Medycznej, Wroclaw
- Romania (7):
  - Spitalui Clinic Judetean de Urgenta, Sectia de Oncologie, Oradea, Bihor County
  - Oncoloab SRL, Craiova, Dolj
  - Centrul de Oncologie Medicala, Iași, Iaşi
  - Institutul Oncologic Al. Trestioreanu Sectia Oncologie Medicala II, Bucharest
  - Institutul Oncologic Al. Trestioreanu, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - Spitalul Clinic Judetean Sibiu, Sibiu
- Russia (10):
  - State Healthcare Institution "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk
  - State Healthcare Institution "Regional Clinical Oncology Dispensary", Kemerovo
  - State Healthcare Institution "Region Clinical Hospital # 1 n.a. professor S.V. Ochapovsky", Krasnodar
  - State Institution "Central Military Clinical Hospital n.a. academician N.N. Burdenko under the Ministry of Defense of Russia", Moscow
  - Institution of the RAMS "Russian Oncology Scientific Centre n.a. N.N. Blokhin under the Russian Academy of Medical Sciences", Moscow
  - State Educational Institution of Higher Professional Education "Saint-Petersburg State Medical University n.a. ac. I.P. Pavlov of the Ministry of Healthcare and Social Development of the Russian Federation", Saint Petersburg
  - Federal State Institution "Petrov Scientific Research Institute of Oncology of Rosmedtechnology", Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "City Clinical Oncology Dispensary", Saint Petersburg
  - Regional State Budget Healthcare Instiution"Tomsk Regional Oncology Dispensary", Tomsk
  - State Healthcare Institution of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
- South Korea (5):
  - Saint Vincent's Hospital, Gyeonggi-do
  - Gachon Medical School Ghil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei Univ. College of Medicine, Seoul
  - Asan Medical Center, Seoul
- Spain (14):
  - ICO (Institut Catalá d´Oncología), L'Hospitalet de Llobregat, Barcelona
  - Fundació Althaia, Manresa, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Oncologico MD Anderson, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario de Valme, Seville
  - Hospital Virgen de la Salud de Toledo, Toledo
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Medical Foundation, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (10):
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Surrey County Hospital NHS Trust, Guildford
  - Leicester Royal Infirmary, Lecester
  - St James' Institute of Oncology, Bexley Wing, St James' University Hospital, Leeds
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Kelly K, Altorki NK, Eberhardt WE, O'Brien ME, Spigel DR, Crino L, Tsai CM, Kim JH, Cho EK, Hoffman PC, Orlov SV, Serwatowski P, Wang J, Foley MA, Horan JD, Shepherd FA. Adjuvant Erlotinib Versus Placebo in Patients With Stage IB-IIIA Non-Small-Cell Lung Cancer (RADIANT): A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2015 Dec 1;33(34):4007-14. doi: 10.1200/JCO.2015.61.8918. Epub 2015 Aug 31. PMID 26324372
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=OSI-774-302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with stage IB to IIIA epidermal growth factor receptor (EGFR)-positive non-small cell lung cancer (NSCLC) were enrolled globally. 1252 patients were enrolled however 2 patients did not have adequate Health Insurance Portability and Accountability Act (HIPAA) documentation and were removed from the database.
Pre-assignment Details: Participants randomized prior to 7 November 2007 comprise the Breached-Protocol Cohort (BPC); those who had not discontinued were offered open-label erlotinib for up to 2 years. Participants randomized subsequently are referred to as the Randomized Cohort.
Groups:
- RC: Erlotinib: Participants in the randomized cohort (RC) who received 150 mg/day erlotinib orally for 2 years or until relapse, death, participant request or investigator decision to discontinue study drug, or intolerable toxicity.
- RC: Placebo: Participants in the randomized cohort (RC) who received matching placebo tablets orally for 2 years or until relapse, death, participant request or investigator decision to discontinue study drug, or intolerable toxicity.
- BPC-NOLC: Erlotinib/Placebo: The BPC no open-label cohort (BPC-NOLC) includes participants randomized prior to 07 November 2007 who did not participate in the open-label erlotinib period and who were previously randomized to receive either erlotinib or placebo in the blinded period, and received at least one dose of erlotinib.
- BPC-NOLC: Placebo Only: The BPC no open-label cohort (BPC-NOLC) includes participants randomized prior to 07 November 2007 who did not participate in the open-label erlotinib period and who were previously randomized to receive either erlotinib or placebo in the blinded period, and did not receive any erlotinib.
- BPC-OLC: Erlotinib: The BPC open-label cohort (BPC-OLC) includes participants randomized prior to 07 November 2007 who received at least 1 dose of study drug after being randomized, who entered the open-label erlotinib period. Data presented for the BPC-OLC included data from both the blinded period and the open-label erlotinib period.
Period: Overall Study
Arm/Group | RC: Erlotinib | RC: Placebo | BPC-NOLC: Erlotinib/Placebo | BPC-NOLC: Placebo Only | BPC-OLC: Erlotinib
Started | 623 | 350 | 134 | 11 | 132
Received Treatment | 612 | 342 | 134 | 7 | 132
Completed | 253 (Completed 2 years of study treatment) | 197 (Completed 2 years of study treatment) | 0 (Completed 2 years of study treatment) | 0 (Completed 2 years of study treatment) | 60 (Completed 2 years of study treatment)
Not Completed | 370 | 153 | 134 | 11 | 72
Not completed — Relapse of NSCLC | 116 | 104 | 19 | 2 | 26
Not completed — Adverse Event | 191 | 22 | 59 | 0 | 34
Not completed — Patient request | 35 | 18 | 43 | 6 | 7
Not completed — Medical/ethical/noncompliance reason | 21 | 9 | 10 | 2 | 5
Not completed — Death | 7 | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RC: Erlotinib | RC: Placebo | BPC-NOLC: Erlotinib/Placebo | BPC-NOLC: Placebo Only | BPC-OLC: Erlotinib | Total
Number analyzed (Participants) | 623 | 350 | 134 | 11 | 132 | 1250
Age, Continuous [Mean (Standard Deviation); unit: years]
  Randomized Cohort | 62.0 (9.28) | 61.8 (9.34) | NA (NA) — Randomized Cohort only | NA (NA) — Randomized Cohort only | NA (NA) — Randomized Cohort only | 61.9 (9.30)
  Breached Protocol Cohort, No Open label | NA (NA) — Breached Protocol Cohort - No Open Label only | NA (NA) — Breached Protocol Cohort - No Open Label only | 64.4 (9.33) | 62.7 (6.23) | NA (NA) — Breached Protocol Cohort - No Open Label only | 64.3 (9.13)
  Breached Protocol Cohort, Open label | NA (NA) — Breached Protocol Cohort - Open Label only | NA (NA) — Breached Protocol Cohort - Open Label only | NA (NA) — Breached Protocol Cohort - Open Label only | NA (NA) — Breached Protocol Cohort - Open Label only | 61.8 (9.35) | 61.8 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 141 | 47 | 2 | 57 | 504
  Male | 366 | 209 | 87 | 9 | 75 | 746
Race/Ethnicity, Customized [Number; unit: participants]
  White | 500 | 279 | 114 | 10 | 111 | 1014
  Black | 14 | 11 | 4 | 0 | 4 | 33
  Asian | 107 | 60 | 15 | 1 | 17 | 200
  American Indian/Alaska Native | 1 | 0 | 1 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 583 | 322 | 123 | 11 | 124 | 1163
  Hispanic or Latino | 40 | 28 | 11 | 0 | 8 | 87
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG criteria: 0: Fully active. 1: Ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of all selfcare. 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours. 4: Completely disabled, no selfcare, totally confined to bed or chair. 5: Dead.
  participants
    Grade 0 | 385 | 211 | 75 | 5 | 77 | 753
    Grade 1 | 230 | 134 | 55 | 6 | 54 | 479
    Grade 2 | 6 | 5 | 3 | 0 | 1 | 15
    Not measured | 2 | 0 | 1 | 0 | 0 | 3
Cigarette Smoking History [Number; unit: participants]
  Never smoked or ≤ 100 cigarettes in lifetime | 129 | 70 | 19 | 1 | 19 | 238
  Former smoker | 423 | 240 | 103 | 9 | 104 | 879
  Current smoker | 71 | 40 | 12 | 1 | 9 | 133
Histology [Number; unit: participants]
  Adenocarcinoma | 367 | 211 | 73 | 3 | 76 | 730
  Squamous cell carcinoma | 196 | 111 | 48 | 8 | 49 | 412
  Undifferentiated large cell | 22 | 8 | 6 | 0 | 4 | 40
  Mixed NSCLC | 29 | 18 | 5 | 0 | 1 | 53
  Other | 9 | 2 | 2 | 0 | 2 | 15
Extent of Disease at Diagnosis [Number; unit: participants] — Staging is based on the size of the main tumor and whether it has grown into nearby areas, the spread of cancer to nearby lymph nodes and whether the cancer has spread (metastasized) to other organs of the body.
  participants
    Stage IA | 1 | 2 | 1 | 0 | 0 | 4
    Stage IB | 329 | 167 | 64 | 4 | 80 | 644
    Stage IIA | 42 | 24 | 10 | 1 | 9 | 86
    Stage IIB | 155 | 99 | 36 | 4 | 23 | 317
    Stage IIIA | 93 | 58 | 21 | 1 | 17 | 190
    Stage IIIB | 2 | 0 | 2 | 0 | 3 | 7
    Stage IV | 1 | 0 | 0 | 1 | 0 | 2
Adjuvant Chemotherapy [Number; unit: participants]
  Yes | 315 | 200 | 63 | 5 | 68 | 651
  No | 308 | 150 | 71 | 6 | 64 | 599
Epidermal Growth Factor Receptor (EGFR) Mutation Status [Number; unit: participants] — EGFR mutation status:
  Activating mutation-positive: exon 19 deletion or exon 21 L858R (or both) detected.
  Wild-type: neither exon 19 deletion nor exon 21 L858R or any other mutation (exon 18, 19, 20 and 21) detected or undetermined.
  Undetermined: exon 19 deletion or exon 21 L858R (or both) mutation status undetermined.
  Activating mutation not positive: neither exon 19 deletion nor exon 21 L858R detected or undetermined (includes other mutation positive and other mutation status undetermined).
  participants
    Activating mutation-positive | 102 | 59 | 10 | 0 | 16 | 187
    Wild-type | 458 | 245 | 116 | 11 | 107 | 937
    Undetermined | 29 | 16 | 1 | 0 | 1 | 47
    Activating mutation not positive | 30 | 27 | 5 | 0 | 6 | 68
    Not Available | 4 | 3 | 2 | 0 | 2 | 11
EGFR Gene Amplification [Number; unit: participants] — Analysis of tumor tissue by fluorescent in situ hybridization (FISH), positivity was defined as amplification (EGFR gene to chromosome ratio of ≥ 2 or ≥ 15 EGFR gene copies in ≥ 10% of tumor cells) or high polysomy (≥ 4 EGFR gene copies in ≥ 40% of tumor cells) .
  participants
    Positive | 445 | 255 | 84 | 8 | 100 | 892
    Negative | 167 | 87 | 49 | 3 | 32 | 338
    Undetermined | 11 | 8 | 1 | 0 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS is the time from the date of randomization until the first day non-small cell lung cancer (NSCLC) relapse is documented by radiological exam and/or biopsy, or until death in the absence of relapse. After randomization, NSCLC relapse was based on radiological evidence or biopsy, as determined by the investigator. Participants without a DFS event were censored on the last adequate radiological assessment date.
Time Frame: Every 3 months during active phase and every 6 months during long term follow-up up to 5 years and yearly thereafter until the data cut-off date of 08 April 2013 (maximum time on follow-up was 64 months).
Population: Randomized cohort full analysis set (all randomized participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 623 | 350
months | 50.5 [44.7 to NA] — Not estimable due to the low number of events | 48.2 [36.0 to NA] — Not estimable due to the low number of events
Statistical Analysis 1: Comparison: Erlotinib vs Placebo; The null hypothesis that DFS distributions of the 2 arms were equivalent was tested using an unstratified 2-sided log-rank test at the 0.05 level. The primary analysis of DFS was performed when at least 410 events had accrued. If the result of the primary analysis of DFS was statistically significant favoring the erlotinib treatment arm, the null hypothesis of no treatment difference of key secondary efficacy variables was tested under a hierarchical testing procedure; Test type: Superiority or Other; p = 0.3235, Log Rank — If the primary analysis of DFS was not statistically significant, the hierarchical testing procedure would stop and all key secondary efficacy analyses would be nonsignificant; any further analysis of these outcomes would be considered exploratory; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.741 to 1.104] — Hazard ratio: erlotinib to placebo

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization until the documented date of death. Participants who were still alive were censored on the last day they were known to be alive.
Time Frame: as for outcome 1
Population: Randomized cohort full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 623 | 350
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

3. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 2
Time Frame: Every 3 months during active phase and every 6 months during long term follow-up up to 5 years and yearly thereafter until the data cut-off date of 11 June 2014 (maximum time on follow-up was 78 months).
Population: Randomized cohort full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 623 | 350
months | NA [77.9 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

4. Secondary Outcome: Disease-free Survival in Participants With EGFR Mutation - Positive Tumors
Description: Disease-free survival (DFS) is the time from the date of randomization until the first day NSCLC relapse is documented by radiological exam and/or biopsy, or until death in the absence of relapse. After randomization, NSCLC relapse was based on radiological evidence or biopsy, as determined by the investigator. Participants without a DFS event were censored on the last adequate radiological assessment date. Activating EGFR mutation-positive is defined as exon 19 deletion or exon 21 L858R (or both) detected.
Time Frame: as for outcome 1
Population: Randomized cohort full analysis set participants who are EGFR mutation positive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 102 | 59
months | 46.4 [39.8 to NA] — Could not be estimated due to low number of events | 28.5 [16.7 to NA] — Could not be estimated due to low number of events

5. Secondary Outcome: Disease-free Survival in Participants With EGFR Mutation - Positive Tumors
Description: as for outcome 4
Time Frame: as for outcome 3
Population: Randomized cohort full analysis set participants who are EGFR mutation positive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 102 | 59
months | 47.8 [39.8 to 60.8] | 28.5 [16.7 to 61.4]

6. Primary Outcome: Disease Free Survival (DFS)
Description: DFS is the time from the date of randomization until the first day that non-small cell lung cancer (NSCLC) relapse is documented by radiological exam and/or biopsy, or until death in the absence of relapse. After randomization, NSCLC relapse was based on radiological evidence or biopsy, as determined by the investigator. Participants without a DFS event were censored on the last adequate radiological assessment date.
Time Frame: Every 3 months during active phase and every 6 months during long term follow-up up to 5 years and yearly thereafter until the data cutoff date of 11 June 2014 (maximum time on follow-up was 78 months).
Population: Randomized cohort full analysis set (all randomized participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 623 | 350
months | 55.0 [47.0 to 64.5] | 56.2 [39.7 to 65.6]
Statistical Analysis 1: Comparison: Erlotinib vs Placebo; The null hypothesis that DFS distributions of the 2 arms were equivalent was tested using an unstratified 2-sided log-rank test at the 0.05 level; Test type: Superiority or Other; p = 0.5620, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.780 to 1.144]

7. Secondary Outcome: Overall Survival in Participants With EGFR Mutation - Positive Tumors
Description: Overall survival is defined as the time from the date of randomization until the documented date of death. Participants who were still alive were censored on the last day they were known to be alive.
  Activating EGFR mutation-positive is defined as exon 19 deletion or exon 21 L858R (or both) detected.
Time Frame: as for outcome 1
Population: Randomized cohort full analysis participants who were EGFR mutation positive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 102 | 59
months | NA [NA to NA] — Could not be estimated due to low number of events | NA [55.4 to NA] — Could not be estimated due to low number of events

8. Secondary Outcome: Overall Survival in Participants With EGFR Mutation - Positive Tumors
Description: as for outcome 7
Time Frame: as for outcome 3
Population: Randomized cohort full analysis participants who were EGFR mutation positive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 102 | 59
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a study participant and did not necessarily have a causal relationship with study treatment.
  An AE was considered serious if it resulted in death, a life-threatening situation, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of a participant, other important medical events, or is on the Astellas Always Serious List.
  A drug-related AE was any AE with at least a possible relationship to study treatment as assessed by the investigator. Severity was graded by the investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events, v3.0, where Grade 1=Mild AE; Grade=2 Moderate AE; Grade 3=Severe AE; Grade 4=Life-threatening or disabling; Grade 5=Death related to AE. AEs leading to death include deaths that occurred more than 30 days after the last dose of study drug.
Time Frame: From the date of first dose of study drug until 30 days after the last dose. The median time on treatment was 11.9 months for erlotinib and 21.9 months for placebo. Data are based off the 11 June 2014 data cut-off date.
Population: Randomized Cohort, safety analysis set: all randomized participants who received at least one dose of study drug. One participant in the Randomized Cohort assigned to the erlotinib arm received placebo instead due to a dispensing error and is included in the placebo group for safety analyses.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 611 | 343
participants
  Any adverse event (AE) | 599 | 307
  Grade 3 or higher adverse event | 279 | 96
  Serious adverse event (SAE) | 118 | 79
  AE leading to discontinuation of study drug | 205 | 29
  AE leading to death | 14 | 5
  AE leading to dose reduction | 150 | 9
  AE leading to dose interruption | 114 | 23
  AE leading to dose interruption and reduction | 156 | 5
  Drug-related AE | 572 | 181
  Drug-related serious AE | 15 | 5
  Drug-related AE leading to discontinuation | 163 | 8

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after the last dose. Maximum time on treatment for the Randomized Cohort was 24 months; maximum time on treatment for the BPC was 13 months on blinded study drug and 26 months on open-label erlotinib.
Description: One participant in the Randomized Cohort assigned to the erlotinib arm received placebo instead due to a dispensing error and is included in the placebo group for safety analyses. For the Breached Protocol Cohort safety analyses are based on the total no open-label and open-label populations.
  Safety data are based on the 11 June 2014 cut-off date.
Arm/Group | RC: Erlotinib | RC: Placebo | BPC-NOLC: Erlotinib/Placebo | BPC-NOLC: Placebo Only | BPC-OLC: Erlotinib
Serious Adverse Events (participants affected / at risk) | 118/611 | 79/343 | 21/134 | 1/11 | 41/132
Other Adverse Events (participants affected / at risk) | 590/611 | 288/343 | 125/134 | 4/11 | 130/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RC: Erlotinib (N=611) | RC: Placebo (N=343) | BPC-NOLC: Erlotinib/Placebo (N=134) | BPC-NOLC: Placebo Only (N=11) | BPC-OLC: Erlotinib (N=132)
Pneumonia (Infections and infestations) | 8 | 2 | 2 | 0 | 3
Respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tooth resorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 3 | 4 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sudden onset of sleep (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Brain mass (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 3
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 0 | 0 | 2
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 3 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Suture rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Cardiovascular insufficiency (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2
Inappropriate affect (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Conjunctival neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RC: Erlotinib (N=611) | RC: Placebo (N=343) | BPC-NOLC: Erlotinib/Placebo (N=134) | BPC-NOLC: Placebo Only (N=11) | BPC-OLC: Erlotinib (N=132)
Rash (Skin and subcutaneous tissue disorders) | 356 | 58 | 51 | 0 | 72
Pruritus (Skin and subcutaneous tissue disorders) | 161 | 51 | 21 | 0 | 29
Dry skin (Skin and subcutaneous tissue disorders) | 127 | 50 | 15 | 0 | 41
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 111 | 19 | 37 | 0 | 45
Alopecia (Skin and subcutaneous tissue disorders) | 67 | 11 | 12 | 0 | 22
Rash erythematous (Skin and subcutaneous tissue disorders) | 30 | 6 | 6 | 0 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 3 | 4 | 0 | 7
Skin fissures (Skin and subcutaneous tissue disorders) | 26 | 2 | 1 | 0 | 9
Acne (Skin and subcutaneous tissue disorders) | 25 | 10 | 6 | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 25 | 5 | 1 | 0 | 7
Erythema (Skin and subcutaneous tissue disorders) | 24 | 5 | 10 | 0 | 13
Nail disorder (Skin and subcutaneous tissue disorders) | 23 | 2 | 1 | 0 | 9
Skin exfoliation (Skin and subcutaneous tissue disorders) | 23 | 4 | 6 | 0 | 8
Exfoliative rash (Skin and subcutaneous tissue disorders) | 19 | 2 | 2 | 0 | 11
Blister (Skin and subcutaneous tissue disorders) | 8 | 0 | 5 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 4 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 10 | 1 | 1 | 1 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 11 | 5 | 0 | 0 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 15 | 4 | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 318 | 54 | 54 | 0 | 86
Nausea (Gastrointestinal disorders) | 84 | 44 | 17 | 1 | 28
Stomatitis (Gastrointestinal disorders) | 61 | 4 | 8 | 0 | 15
Vomiting (Gastrointestinal disorders) | 55 | 23 | 10 | 0 | 12
Constipation (Gastrointestinal disorders) | 35 | 23 | 7 | 0 | 14
Abdominal pain (Gastrointestinal disorders) | 34 | 11 | 6 | 0 | 14
Dyspepsia (Gastrointestinal disorders) | 30 | 14 | 4 | 0 | 15
Abdominal pain upper (Gastrointestinal disorders) | 28 | 20 | 0 | 0 | 11
Dry mouth (Gastrointestinal disorders) | 21 | 3 | 7 | 0 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 20 | 8 | 1 | 0 | 4
Cheilitis (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 8
Mouth ulceration (Gastrointestinal disorders) | 13 | 1 | 1 | 0 | 5
Flatulence (Gastrointestinal disorders) | 11 | 6 | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 121 | 69 | 17 | 0 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 85 | 61 | 15 | 0 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47 | 4 | 4 | 0 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 | 4 | 3 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12 | 3 | 0 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 3 | 0 | 6
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 3 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 2 | 0 | 4
Fatigue (General disorders) | 118 | 49 | 23 | 0 | 34
Asthenia (General disorders) | 37 | 21 | 6 | 0 | 6
Mucosal inflammation (General disorders) | 27 | 2 | 6 | 0 | 12
Pyrexia (General disorders) | 23 | 13 | 6 | 1 | 9
Xerosis (General disorders) | 19 | 5 | 0 | 0 | 1
Oedema peripheral (General disorders) | 18 | 11 | 1 | 0 | 5
Chest pain (General disorders) | 15 | 12 | 2 | 0 | 4
Non-cardiac chest pain (General disorders) | 12 | 9 | 1 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 40 | 24 | 3 | 0 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 36 | 7 | 1 | 0 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 28 | 10 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 25 | 4 | 0 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 12 | 3 | 0 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 23 | 2 | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 6 | 4 | 0 | 6
Paronychia (Infections and infestations) | 39 | 2 | 4 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 30 | 15 | 0 | 0 | 13
Nasopharyngitis (Infections and infestations) | 29 | 30 | 2 | 0 | 17
Bronchitis (Infections and infestations) | 21 | 12 | 1 | 0 | 9
Rash pustular (Infections and infestations) | 19 | 1 | 3 | 0 | 13
Urinary tract infection (Infections and infestations) | 19 | 12 | 1 | 0 | 3
Sinusitis (Infections and infestations) | 7 | 8 | 3 | 0 | 7
Ear infection (Infections and infestations) | 2 | 1 | 0 | 0 | 5
Nail infection (Infections and infestations) | 2 | 0 | 1 | 0 | 5
Rhinitis (Infections and infestations) | 12 | 6 | 1 | 0 | 5
Localised infection (Infections and infestations) | 4 | 2 | 0 | 0 | 4
Pneumonia (Infections and infestations) | 16 | 5 | 1 | 0 | 4
Skin infection (Infections and infestations) | 3 | 0 | 1 | 0 | 4
Headache (Nervous system disorders) | 42 | 40 | 10 | 0 | 13
Dizziness (Nervous system disorders) | 26 | 22 | 9 | 1 | 13
Dysgeusia (Nervous system disorders) | 26 | 4 | 5 | 0 | 13
Paraesthesia (Nervous system disorders) | 20 | 15 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 4 | 0 | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 9 | 2 | 1 | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 4 | 2 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 80 | 24 | 20 | 1 | 20
Dehydration (Metabolism and nutrition disorders) | 5 | 1 | 4 | 0 | 4
Insomnia (Psychiatric disorders) | 40 | 21 | 6 | 0 | 16
Depression (Psychiatric disorders) | 33 | 12 | 5 | 0 | 6
Anxiety (Psychiatric disorders) | 20 | 14 | 5 | 0 | 7
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 56 | 19 | 2 | 0 | 19
Weight increased (Investigations) | 16 | 20 | 1 | 0 | 6
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 6 | 1 | 0 | 4
Conjunctivitis (Eye disorders) | 34 | 0 | 1 | 0 | 5
Dry eye (Eye disorders) | 31 | 3 | 6 | 0 | 5
Hypertension (Vascular disorders) | 22 | 14 | 2 | 0 | 8
Eye irritation (Eye disorders) | 8 | 3 | 2 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 9 | 6 | 4 | 0 | 5
Anaemia (Blood and lymphatic system disorders) | 16 | 6 | 2 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 6 | 6 | 1 | 0 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 18 | 7 | 2 | 0 | 8

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the currency or completeness of the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 60 days prior to publication for review and comment. Sponsor may delay the publication for up to 6 months to seek patent protection.